CLINICAL TRIAL: NCT01114763
Title: Hämeenlinna Metabolic Syndrome Research Program (HMS): Comparison of Men With Metabolic Syndrome and Their Physically Active Controls - Circulating Oxidized LDL and Arterial Elasticity
Brief Title: Hämeenlinna Metabolic Syndrome Research Program: Oxidized LDL and Arterial Elasticity in Metabolic Syndrome and Controls (HMS-01)
Acronym: HMS-01
Status: Completed | Type: Observational
Sponsor: Kanta-Häme Central Hospital (Other Government)
Collaborators: Linnan Klinikka Oy (Other)
Responsible Party: Ari Palomäki, MD PhD, Head of department, Central Hospital of Kanta-Häme, Hämeenlinna, Finland
Other Study IDs: KHMetS-01-AP
Record Dates: First submitted 2010-04-30; First posted 2010-05-03 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-04

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Oxidized Low Density Lipoprotein; Arterial Elasticity; Diabetes Mellitus; Cardiovascular Diseases
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum, EDTA plasma, citrate plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Metabolic syndrome: 40 men with metabolic syndrome
- Control: 40 physically active men

SUMMARY:
Mechanisms that link metabolic syndrome to atherosclerosis are incompletely understood. As a part of Hämeenlinna Metabolic Syndrome Research Program (HMS), 40 men with metabolic syndrome and their 40 physically active controls (age: 30 to 65 years) are compared in a cross-sectional study. Except routine laboratory parameters, arterial elasticity and levels of oxidized LDL are determined.

Study hypothesis: Levels of oxidized LDL and findings in arterial elasticity may differ between subjects with metabolic syndrome and controls explaining the elevated risk for cardiovascular diseases among patients with metabolic syndrome.

DETAILED DESCRIPTION:
Accumulation of oxidized low-density lipoproteins in the intimae of arteries together with risk factors known to enhance atherosclerosis, damage the endothelium of the arterial wall. Dysfunction of the endothelium leads into loss of elasticity of the artery. Especially a reduction in the elasticity of small arteries has been found prominent in atherosclerosis and is believed to serve as a marker for early stages of atherosclerosis.

In this study, we investigate whether the levels of oxidized LDL and arterial elasticity differ between patients with metabolic syndrome and their physically active controls. Oxidized LDL is assessed by a two-site ELISA immunoassay (Mercodia, Uppsala, Sweden). The capacitive elasticity of large arteries (C1) and the reflective elasticity of small arteries (C2) are automatically assessed by the CR-2000 as a mean of five most similar pulse waves appearing during the measurement. C1 identifies the elastic properties of aorta and other large arteries, C2 the endothelial function of the microvascular circulation. Proper statistical methods are used to reveal possible differences and their significance between the patients and controls.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Metabolic syndrome

* 40 Finnish men with metabolic syndrome (MetS) defined according to National Cholesterol Education Program (NCEP) Adult Treatment Panel III
* MetS diagnosed in routine health examination and laboratory tests
* Age: 30 to 65 years

Group 2: Control

* 40 age-matched men
* Exercise physically more than three times a week and more than 30 minutes per exercise on regular basis
* Never been studied or treated because of cardiovascular disease

Exclusion Criteria:

* Cholesterol-lowering medication
* ACE-inhibitor medication
* Angiotensin-receptor blocker medication

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2003-06; Primary Completion 2005-11 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari K Palomäki, MD PhD, Study Director — Central Hospital of Kanta-Häme; Kalevi Oksanen, MD PhD, Study Director — Central Hospital of Kanta-Häme
Locations (2):
- Finland (2):
  - Linnan Klinikka, Hämeenlinna
  - Central Hospital of Kanta-Häme, Hämeenlinna

REFERENCES:
- [Derived] Pohjantahti-Maaroos H, Palomaki A, Kankkunen P, Laitinen R, Husgafvel S, Oksanen K. Circulating oxidized low-density lipoproteins and arterial elasticity: comparison between men with metabolic syndrome and physically active counterparts. Cardiovasc Diabetol. 2010 Aug 20;9:41. doi: 10.1186/1475-2840-9-41. PMID 20727144